CLINICAL TRIAL: NCT01503359
Title: Effect of Sarcosine on Symptomatology, Quality of Life, Cognitive and Sexual Functioning, Blood Levels of Sarcosine, Glycine, BDNF and MMP-9, Oculomotor, Brain Metabolism and Oxidative Stress Parameters in Schizophrenia.
Brief Title: Effect of Sarcosine on Symptomatology, Quality of Life, Oxidative Stress and Glutamatergic Parameters in Schizophrenia
Acronym: PULSAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Dominik Strzelecki MD PhD, Principal Investigator, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PULSAR; N N402 268836 (Other Grant/Funding Number: Ministry of Science and Higher Education, Poland)
Record Dates: First submitted 2011-12-30; First posted 2012-01-04 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Schizophrenia
Keywords: glutamic acid; sarcosine; NMDA; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Sarcosine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Supplement: Sarcosine (Experimental): Sarcosine Group
  Interventions: Dietary Supplement: Sarcosine
- Placebo (Placebo Comparator): Control Group
  Interventions: Dietary Supplement: Sarcosine

INTERVENTIONS:
Dietary Supplement: Sarcosine — Sarcosine group patients will receive 2 grams of sarcosine once a day in the morning for 6 months.
  Placebo group patients will receive 2 grams of placebo once a day in the morning for 6 months.
  Other Names: glycine transporter inhibitor; GlyT1 inhibitor

SUMMARY:
The purpose of study is to determine whether dietary supplement sarcosine is effective in treatment of schizophrenia. The investigators will assess impact of sarcosine on quality of life and sexual functioning. In this project the investigators will also measure glycine, sarcosine, BDNF, MMP-9 levels and oxydative stress parameters in blood, brain glutamatergic metabolism parameters in magnetic resonance spectroscopy and oculomotoric changes in electrooculography.

DETAILED DESCRIPTION:
Glutamic acid is the largest excitatory neurotransmitter in the central nervous system, the population of glutamatergic neurones represents approximately 50% of all neurones in the brain. Being closely dependent on the inhibitory GABA system, the glutamate system is responsible for the transmission and modulation of the majority of brain signals and connected with dopaminergic and serotonergic systems. The glutamate system plays an important role in the pathogenesis of schizophrenia. NMDA receptor antagonists, including phencyclidine, ketamine and MK-801, cause symptoms similar to those found in schizophrenia, as well as deterioration of mental state in patients with schizophrenia. What is important from a theoretical point of view NMDA agonists also cause negative symptoms which are not observed after amphetamine or other drugs intoxications. Based on these observations, it was assumed that normalization of glutamatergic transmission may result in an improvement in schizophrenia symptomatology.

According to the assumptions of this hypothesis, attempts were made to stimulate transmission within this system. Due to the high risk of excitotoxic effects induction therapy with glutamic acid is not administered (hyperactivity of glutamatergic system, leading to nerve cell damage was observed in neurodegenerative diseases). Along with glutamic acid and voltage changes dependent on another glutamatergic receptor - AMPA, presence of glycine is necessary to stimulate the NMDA receptor. This widely distributed amino acid, an important element of protein chains, is present in a daily diet (average consumption amounts to 2g/day). In addition to building properties, it is of paramount importance in the central nervous system. As a primary transmitter in glycinergic neurones it belongs to the class I of neurotransmitters. Moreover, it also plays a role as a co-agonist and a modulator, for example in the glutamatergic system. Glutamic acid is released from nerve endings into the synaptic cleft, where it is re-uptaken and dispersed, which, in consequence, results in a rapid decline in its concentration in the vicinity of NMDA receptors. As a result, the time of receptor binding is short. Intrasynaptic glycine turnover is different - it resides inside the synapses permanently, depending on the concentration and, to a greater or lesser extent, binds to a modulatory site. Glial cells, with identified glycine transport system (GlyT-1) are responsible for maintaining a stable level of glycine in neuronal junctions. New research on inhibitors of this transport system (GTI) eg. sarcosine, which may have similar or better effects to glycine administration, have begun. Glycine does not bind to all the modulatory sites on NMDA receptor in vivo, and augmentation of this saturation intensifies glutamatergic transmission. This phenomenon is particularly observed in individuals with relatively low (not sufficient for maximum saturation of the receptor site) levels of synaptic glycine.

We hypothesize that supplementation of sarcosine helps achieve betterment in symptomatology, general quality of life and also cognitive functioning and other prefrontal derivatives, eg. oculomotor functions.

To extend research we planned assessing blood levels of glycine, sarcosine but also other parameters involved in glutamatergic transmission such as BDNF and metalproteinase MMP-9. Knowing excitotoxic properties of glutamate TBARS (thiobarbituric acid reactive substances) - oxidative stress related will be assessed.

Methodology of the study. We plan to enroll 60-70 patients in stable mental state meeting criteria for schizophrenia according to ICD-10 with predominant negative symptoms (minimum of 21 points and severity of each negative symptom at least 3 points in PANSS-Negative subscale).

Main study part will be continued for 26 weeks (T0-T26) and 10 visits (W1-W10). The preceding 12-week period (W0-W1) will be used for evaluation of stability of mental state and pharmacotherapy.

Patients on visit T0 will be randomized to two comparable groups of 30 patients (sarcosine and control group). Researchers and patients will not have information on the administered treatment.

During the study patients will receive previous antipsychotic treatment (at least 3-month without dosage change). Mental stability will be assessed during the preceding period (W1 and W0 visit - 12 weeks before W1). Sarcosine (or placebo) will be augmented between visits W1 and W9, the subsequent period (between W9 and W10), will be used to evaluate the consequences of withdrawal sarcosine (and placebo).

Information on the history of the disease, and current mental status will be obtained during the psychiatric examination, in part, standardized by the use of commonly accepted psychiatric scales (PANSS, Calgary Depression Scale, CGI, SAS and quality of life and sexual activity scales). Assessment of the use of psychiatric scales will be used on each of the visits.

As the basic tools used to study cognitive functioning test Wisconsin Card Sorting (WCST), Trail Making Test (TMT) and Stroop Test will be used. Psychological testing will be performed by a psychologist on visits W1, W6 and W9.

Assessment of metabolism of glycine and glutamic acid in brain tissue in the frontal cortex and hippocampus using magnetic resonance spectroscopy, electrooculography, parameter of oxidative stress - T-BARS and blood assessments (glycine, sarcosine, BDNF and MMP-9) will be performed on visits W1 and W9.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of schizophrenia (ICD-10)

Other criteria related to the diagnosis verified during the selection visit:

* The score for the PANSS negative symptoms subscale ≥ 21,
* Severity of individual symptoms in the PANSS positive symptoms subscale may not exceed 3 points.

Exclusion Criteria:

General

* lack of written informed consent,
* risk of noncompliance during the study period,
* patients who can not be assessed throughout the study period (eg. due to travel or vacations),
* pregnancy or breastfeeding,
* women of childbearing potential not using effective contraception (ie. birth control pill, surgical sterilization, hormonal contraceptive injection, IUD, contraceptive implant, patch, or condoms),
* participation in another clinical study, currently or within 3 months before the visit of a selection panel
* patients previously subjected to selection for this study.

Medical and Therapeutic Criteria Associated with schizophrenia

* patients in acute psychosis, severe symptoms of productive,
* patients taking clozapine,
* declaring suicidal tendencies, history of committing suicide in the past year.

Associated with other psychiatric disorders

* patients currently meeting criteria for ICD-10 diagnosis of mental disorder other than schizophrenia (in the last 6 months before the visit of a selection), confirmed by the MINI questionnaire
* patients showing a prevalent and / or severe symptoms of depression (even without meeting criteria for major depressive episode according to ICD-10 criteria),
* patients ever diagnosed with lifetime bipolar disorder,
* patients with severe personality disorders, particularly type of antisocial, borderline, or histrionicznego that could affect the assessment of test results.

Other

* abuse or addiction to alcohol or psychoactive substances (excluding nicotine) within the last 6 months, according to the criteria of ICD-10, confirmed by the MINI questionnaire,
* disturbances occurring in the form of somatic according to ICD-10 criteria,
* Delirium or dementia according to ICD-10 criteria,
* current diagnosis of neurological diseases (eg, stroke, seizures, migraine, multiple sclerosis),
* liver failure (ie, cirrhosis or active liver disease), diagnosed acute or chronic hepatitis,
* severe or uncontrolled somatic disease that could affect the course of the study (eg cancer, cardiovascular, respiratory, metabolic or oral, severe renal failure, unstable diabetes type I or II, morbid obesity, untreated or uncontrolled hypertension, clinically significant blood),
* thyroid dysfunction (especially hypothyroidism) untreated or uncontrolled, T - thyroid hormones treatment started, terminated or modified in the 3 months before the selection visit,
* hormone replacement therapy started, terminated or modified in the 3 months before the selection visit.
* recognized disorders of hemostasis,

Associated with a prior or concomitant treatment Particular caution should be maintained when using drugs likely to affect the central nervous system - their mechanism of action could affect the course of the study. Use of these substances after the selection visit is not allowed.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-02 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Assessment of sarcosine vs. placebo impact on schizophrenia symptoms using Positive and Negative Syndrome Scale (PANSS). | 6 months
  Both arms, every visit

SECONDARY OUTCOMES:
Impact assessment of sarcosine versus placebo on the parameters of quality of life (QoL) and sexual functioning. | 6 months
  Both arms, every visit
Impact assessment of sarcosine versus placebo on depressive symptoms using Calgary Depression Scale for Schizophrenia. | 6 months
  Both arms, every visit
Impact assessment of sarcosine versus placebo on cognitive functions using Wisconsin Card Sort Test, Trail Making Test and Stroop Test. | 6 months
  Both arms, before and after taking sarcosine or placebo
Impact assessment of sarcosine versus placebo on oxidative stress parameters (T-BARS). | 6 months
  Both arms, before and after taking sarcosine or placebo
Impact assessment of sarcosine versus placebo on brain metabolism parameters (magnetic resonance spectroscopy). | 6 months
  Both arms, before and after taking sarcosine or placebo
Impact assessment of sarcosine versus placebo on oculomotoric parameters (saccadic and antisaccadic task in electrooculography). | 6 months
  Both arms, before and after taking sarcosine or placebo
Impact assessment of sarcosine versus placebo on blood levels of glycine, sarcosine, BDNF and MMP-9. | 6 months
  Both arms, before and after taking sarcosine or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Strzelecki, MD, PhD, Principal Investigator — Department of Affective and Psychotic Disorders, Medical University of Lodz; Jolanta Rabe-Jabłońska, MD, PhD, Study Chair — Department of Affective and Psychotic Disorders, Medical University of Lodz
Locations (1):
- Central Clinical Hospital, Lodz, Czechosłowacka 8/10, Poland

REFERENCES:
- [Background] Carlsson A, Waters N, Waters S, Carlsson ML. Network interactions in schizophrenia - therapeutic implications. Brain Res Brain Res Rev. 2000 Mar;31(2-3):342-9. doi: 10.1016/s0165-0173(99)00050-8. PMID 10719161
- [Background] Carlsson M, Carlsson A. Interactions between glutamatergic and monoaminergic systems within the basal ganglia--implications for schizophrenia and Parkinson's disease. Trends Neurosci. 1990 Jul;13(7):272-6. doi: 10.1016/0166-2236(90)90108-m. PMID 1695402
- [Background] Coyle JT. The glutamatergic dysfunction hypothesis for schizophrenia. Harv Rev Psychiatry. 1996 Jan-Feb;3(5):241-53. doi: 10.3109/10673229609017192. PMID 9384954
- [Background] Gao XM, Sakai K, Roberts RC, Conley RR, Dean B, Tamminga CA. Ionotropic glutamate receptors and expression of N-methyl-D-aspartate receptor subunits in subregions of human hippocampus: effects of schizophrenia. Am J Psychiatry. 2000 Jul;157(7):1141-9. doi: 10.1176/appi.ajp.157.7.1141. PMID 10873924
- [Background] Goff DC, Herz L, Posever T, Shih V, Tsai G, Henderson DC, Freudenreich O, Evins AE, Yovel I, Zhang H, Schoenfeld D. A six-month, placebo-controlled trial of D-cycloserine co-administered with conventional antipsychotics in schizophrenia patients. Psychopharmacology (Berl). 2005 Apr;179(1):144-50. doi: 10.1007/s00213-004-2032-2. Epub 2004 Oct 21. PMID 15502972
- [Background] Goff DC, Coyle JT. The emerging role of glutamate in the pathophysiology and treatment of schizophrenia. Am J Psychiatry. 2001 Sep;158(9):1367-77. doi: 10.1176/appi.ajp.158.9.1367. PMID 11532718
- [Background] Javitt DC, Silipo G, Cienfuegos A, Shelley AM, Bark N, Park M, Lindenmayer JP, Suckow R, Zukin SR. Adjunctive high-dose glycine in the treatment of schizophrenia. Int J Neuropsychopharmacol. 2001 Dec;4(4):385-91. doi: 10.1017/S1461145701002590. PMID 11806864
- [Background] Javitt DC, Zukin SR. Recent advances in the phencyclidine model of schizophrenia. Am J Psychiatry. 1991 Oct;148(10):1301-8. doi: 10.1176/ajp.148.10.1301. PMID 1654746
- [Background] Lane HY, Liu YC, Huang CL, Chang YC, Liau CH, Perng CH, Tsai GE. Sarcosine (N-methylglycine) treatment for acute schizophrenia: a randomized, double-blind study. Biol Psychiatry. 2008 Jan 1;63(1):9-12. doi: 10.1016/j.biopsych.2007.04.038. Epub 2007 Jul 20. PMID 17659263
- [Background] Lane HY, Huang CL, Wu PL, Liu YC, Chang YC, Lin PY, Chen PW, Tsai G. Glycine transporter I inhibitor, N-methylglycine (sarcosine), added to clozapine for the treatment of schizophrenia. Biol Psychiatry. 2006 Sep 15;60(6):645-9. doi: 10.1016/j.biopsych.2006.04.005. Epub 2006 Jun 14. PMID 16780811
- [Background] Law AJ, Deakin JF. Asymmetrical reductions of hippocampal NMDAR1 glutamate receptor mRNA in the psychoses. Neuroreport. 2001 Sep 17;12(13):2971-4. doi: 10.1097/00001756-200109170-00043. PMID 11588613
- [Background] McBain CJ, Mayer ML. N-methyl-D-aspartic acid receptor structure and function. Physiol Rev. 1994 Jul;74(3):723-60. doi: 10.1152/physrev.1994.74.3.723. No abstract available. PMID 8036251
- [Background] Olney JW, Newcomer JW, Farber NB. NMDA receptor hypofunction model of schizophrenia. J Psychiatr Res. 1999 Nov-Dec;33(6):523-33. doi: 10.1016/s0022-3956(99)00029-1. PMID 10628529
- [Background] Tsai G, Lane HY, Yang P, Chong MY, Lange N. Glycine transporter I inhibitor, N-methylglycine (sarcosine), added to antipsychotics for the treatment of schizophrenia. Biol Psychiatry. 2004 Mar 1;55(5):452-6. doi: 10.1016/j.biopsych.2003.09.012. PMID 15023571
- [Background] Tsai G, van Kammen DP, Chen S, Kelley ME, Grier A, Coyle JT. Glutamatergic neurotransmission involves structural and clinical deficits of schizophrenia. Biol Psychiatry. 1998 Oct 15;44(8):667-74. doi: 10.1016/s0006-3223(98)00151-6. PMID 9798069
- [Background] Tuominen HJ, Tiihonen J, Wahlbeck K. Glutamatergic drugs for schizophrenia. Cochrane Database Syst Rev. 2006 Apr 19;2006(2):CD003730. doi: 10.1002/14651858.CD003730.pub2. PMID 16625590
- [Background] West AR, Floresco SB, Charara A, Rosenkranz JA, Grace AA. Electrophysiological interactions between striatal glutamatergic and dopaminergic systems. Ann N Y Acad Sci. 2003 Nov;1003:53-74. doi: 10.1196/annals.1300.004. PMID 14684435
- [Background] Yurgelun-Todd DA, Coyle JT, Gruber SA, Renshaw PF, Silveri MM, Amico E, Cohen B, Goff DC. Functional magnetic resonance imaging studies of schizophrenic patients during word production: effects of D-cycloserine. Psychiatry Res. 2005 Jan 30;138(1):23-31. doi: 10.1016/j.pscychresns.2004.11.006. PMID 15708298
- [Background] Zafra F, Aragon C, Olivares L, Danbolt NC, Gimenez C, Storm-Mathisen J. Glycine transporters are differentially expressed among CNS cells. J Neurosci. 1995 May;15(5 Pt 2):3952-69. doi: 10.1523/JNEUROSCI.15-05-03952.1995. PMID 7751957
- [Derived] Strzelecki D, Podgorski M, Kaluzynska O, Stefanczyk L, Kotlicka-Antczak M, Gmitrowicz A, Grzelak P. Adding Sarcosine to Antipsychotic Treatment in Patients with Stable Schizophrenia Changes the Concentrations of Neuronal and Glial Metabolites in the Left Dorsolateral Prefrontal Cortex. Int J Mol Sci. 2015 Oct 15;16(10):24475-89. doi: 10.3390/ijms161024475. PMID 26501260
- [Derived] Strzelecki D, Podgorski M, Kaluzynska O, Gawlik-Kotelnicka O, Stefanczyk L, Kotlicka-Antczak M, Gmitrowicz A, Grzelak P. Supplementation of antipsychotic treatment with sarcosine - GlyT1 inhibitor - causes changes of glutamatergic (1)NMR spectroscopy parameters in the left hippocampus in patients with stable schizophrenia. Neurosci Lett. 2015 Oct 8;606:7-12. doi: 10.1016/j.neulet.2015.08.039. Epub 2015 Aug 22. PMID 26306650